CLINICAL TRIAL: NCT02786888
Title: Prospective Comparison of Adductor Canal Block Performed With a Multiport Versus Single Bevel Needle
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeff Swenson, M.D., University of Utah
Other Study IDs: IRB 00090426
Record Dates: First submitted 2016-05-17; First posted 2016-06-01 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- conventional needle: conventional needle used
- fenestrated needle: fenestrated needle used

SUMMARY:
Early ambulation after knee replacement surgery is made possible in large part by providing safe and effective pain control. Peripheral nerve blocks are increasingly used for postoperative analgesia since they can provide excellent pain relief and minimize the need for opioid analgesics.

Ultrasound guided adductor canal block (ACB) was first reported in 2009 by anesthesiologists at the University of Utah. This block is unique in that it spares motor function in the lower extremity. Since 2009, a number of publications have described the successful use of ACB for pain management after total knee arthroplasty (TKA), anterior cruciate ligament (ACL) reconstruction, and other procedures of the knee. As a component of multi-modal analgesia, ACB can provide effective postoperative pain control and facilitate early hospital discharge.

Although it is widely utilized, the ACB block can be technically difficult to perform since it requires injection in immediate proximity to the femoral artery and vein. In patients with a large thigh circumference, ultrasound can be challenging since the femoral vessels are deeper and more difficult to visualize. This presents the possibility of vessel trauma and/or intravascular injection of local anesthetic.

The investigators have implemented a new technique for performing the ACB. This block is performed using a 20G fenestrated needle. The needle is FDA approved for peripheral nerve block. It has an occluded tip with 8 side ports on alternating sides of the distal 2cm. Injection through the fenestrated needle produces effective distribution of local anesthetic to nerves of the adductor canal without immediate proximity to the femoral artery and vein. The ultrasound landmarks used to perform ACB with the fenestrated needle are readily visible even in patients with very large thigh circumference.

In summary, early experience with the US guided ACB block performed with a fenestrated block needle suggests that it is technically easier and potentially safer to perform than blocks performed with a conventional needle.

This study should be performed prospectively in order to ensure accurate data comparing the two needles. A retrospective review of blocks performed using a conventional needle would not provide accurate data with respect to the number of attempts, time required to perform the blocks or the resulting sensory changes after performing the nerve block.

DETAILED DESCRIPTION:
A new fenestrated (multiple side-ports) needle has recently been cleared by the FDA for performing peripheral nerve blocks. Experience with this needle suggests that it can make ACB technically easier and safer to perform.This is due in large part because it eliminates the need to position the needle in close proximity to large blood vessels in the thigh.

The objectives for this study would be to prospectively compare nerve blocks performed for postoperative analgesia performed using conventional (single bevel) needles to those performed using the fenestrated needle. Specifically, the investigators would compare metrics such as; time to perform the block, number of attempts, unintentional blood vessel puncture, and successful injection rates. Successful injection rates would be quantified by comparing the distribution of sensory loss after each injection. Those injections resulting in a loss of sensation over the skin surfaces innervated by nerves of the adductor canal would be judged to be "successful". An absence of sensory change in these surfaces would be judged as "unsuccessful".

Procedures:

All patients will be randomized to receive treatment with one of two nerve block needles. Neither the investigators nor the patients will be blinded. Randomization will be based solely on the results of a computer generated random sequence.

All patients participating in the study will receive the same anesthetic, surgery, postoperative care, and pain management that is provided currently for patients (including those not enrolled in this study protocol) having knee replacement at the University of Utah. This investigation is designed to compare only the efficacy of two needle designs that are currently used and FDA approved for peripheral nerve block.

Patients consenting to participate in the study will be randomized to receive an ACB performed with either a single bevel (conventional) or a fenestrated needle. The ACB will be placed in the preoperative holding area approximately 30 minutes before being transported to the operating room. During performance of the nerve block, the time to complete the nerve block, the number of attempts used to complete the nerve block, the incidence of blood vessel puncture and/or blood aspiration will be recorded for each case. All patients will also be assessed for sensory changes in the lower extremity as a metric for block efficacy.

In the operating room, patients will be anesthetized using a spinal block and will receive intravenous sedation at the discretion of the attending anesthesiologist.

During the postoperative period, the quality and duration of analgesia will be primary metrics used to compare the two study needles. Specifically, numerical pain scores reported by the patients and opioid consumption will be compared for both groups.

All patients for whom the is a possible "failed nerve block" will be offered a repeat "rescue" nerve block after surgery. A failed block would be defined by an absence of sensory changes in the extremity associated with poor pain control reported by the patient.

Additional metrics for comparison would be the time to ambulation after surgery and the time to hospital discharge.

Statistical Methods, Data Analysis and Interpretation

The study will be prospective and randomized for two groups of patients having nerve blocks as part of their pain management protocol for total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* all TKA patients

Exclusion Criteria:

* refuse nerve block

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients for elective knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
The efficiency in performing nerve block | this metric will be obtained while the nerve block is being performed
  The number of attempts during block placement as well as the number of times the needle must be repositioned during block placement. This will simply be recorded as a whole number by the study nurse. The number of unintended vascular punctures observed by a study nurse will be recorded.

SECONDARY OUTCOMES:
pain control as a measure of nerve block effectiveness will be recorded using a verbal analog scale between 1 and 10. Opioid requirements will be recorded as a total number of milligrams received. | this metric will be recorded during the first 24 hours after surgery
  the pain scores and opioid requirements resulting after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Swenson, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swenson JD, Pollard JE, Peters CL, Anderson MB, Pace NL. Randomized controlled trial of a simplified adductor canal block performed for analgesia following total knee arthroplasty. Reg Anesth Pain Med. 2019 Mar;44(3):348-353. doi: 10.1136/rapm-2018-100070. Epub 2019 Jan 23. PMID 30679333